CLINICAL TRIAL: NCT00600678
Title: Characterisation of Gastric Emptying of a High Caloric Sip Feed Using the Paracetamol Absorption Method: Intraindividual Comparison of Paracetamol Pharmacokinetics After Oral co-Administration With Sip-Feed and After Intravenous Administration in Healthy Volunteers of Both Genders in an Open, Single Centre Study
Brief Title: Gastric Emptying Study After Administration of a High Caloric Sip Feed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Frank Folchert, Fresenius Kabi Deutschland GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N-PRX-02-DE
Record Dates: First submitted 2008-01-07; First posted 2008-01-25 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Enteral Nutrition
Keywords: food for special medical purposes
MeSH Terms: interventions — Dietary Supplements; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: ProvideXtra DRINK (oral nutritional supplement, food for special medical purposes)

INTERVENTIONS:
Dietary Supplement: ProvideXtra DRINK (oral nutritional supplement, food for special medical purposes) — Single, oral administration of nutritional supplement under fasting condition within 2 minutes.

SUMMARY:
Measurement of gastric emptying time of an oral nutritional supplement (ProvideXtra DRINK) by using the paracetamol absorption method in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* caucasian origin
* BMI: 22kg/m2 - 27kg/m2;

Exclusion Criteria:

* existing diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of paracetamol (e.g. gastrointestinal or liver disease),
* known allergic reactions to investigational products,
* diseases and/or pathological findings, which could affect absorption, metabolism and/or gastric emptying (e.g. dyspepsia and gastroesophageal reflux),
* regular medication which can influence hepatic biotransformation and/or absorption,
* alcohol dependence, blood donation;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
- Gastric emptying after a single oral administration of a nutritional supplement | Time frame gastric emptying: blood samples will be taken at predefined time points, up to 12h after application of test product.

SECONDARY OUTCOMES:
safety and tolerability | entire study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Germany
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany